CLINICAL TRIAL: NCT01907295
Title: National Cohort Study of Idiopathic and Heritable Pulmonary Arterial Hypertension
Acronym: NAIAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Collaborators: British Heart Foundation (Other); Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Nick Morrell, BHF Professor of Cardiopulmonary Medicine, University of Cambridge
Other Study IDs: A092860
Record Dates: First submitted 2013-07-08; First posted 2013-07-24 (Estimated); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: idiopathic; heritable; anorexigen; PCH/PVOD
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — All subjects will have a sample of blood taken for next generation genetic sequencing (up to their entire genome). Samples will be sequenced to identify novel genetic mutations associated with PAH. This blood sample will be taken once during the study
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients: Patients diagnosed with idiopathic, anorexigen-induced, heritable PAH and PVOD/PCH
- Relatives and controls: Relative has a family member diagnosed with idiopathic, anorexigen-induced, heritable PAH and PVOD/PCH Self declared healthy individuals

SUMMARY:
Pulmonary arterial hypertension (PAH), or high blood pressure in the lungs, is a rare condition that can shorten life. Although the cause of this disease is usually unknown, in about 70% of heritable and 15-20% of idiopathic cases there is a change in a gene (a mutation) that controls how blood vessels grow and function. The gene is called bone morphogenetic protein type receptor 2 (BMPR2). Although mutations in BMPR2 are a risk factor for PAH, not everyone with a mutation gets the disease. Additional genetic and environmental factors are likely to contribute. The investigators suspect that mutations in other genes are responsible for some cases of PAH. In this study the investigators aim to recruit all patients with PAH and some of their relatives and follow them up for several years. The investigators hope to discover new mutations for this disease and to determine what factors lead to poor outcome, and to understand what triggers disease in patients with mutations.

Who can participate? Adults with PAH, their relatives and controls (one off blood sample)

DETAILED DESCRIPTION:
What does the study involve?

PAH patients will be seen at their local centre by their service team but they will have additional bloods taken. Relatives of PAH patients will be seen every year at their nearest PAH centre. Tests will include:

* Epidemiology Questionnaire to assess factors affecting health
* An echocardiogram (ECHO) to assess the size, shape, pumping action and the extent of any damage to the heart.
* Lung function tests which include blowing measurements to assess gas volumes within the lungs as well as assessment of how the lungs exchange gases.
* Optional right heart catheterisation (RHC) to determine how much blood your heart is pumping while you are resting and on exercise. Optional Cardiac Magnetic Resonance tests. To measure heart function. ( to be done only once)
* 6 minute walk test. To measure exercise capacity
* Cardiopulmonary exercise test. A bicycle exercise test, which will indicate how much blood your heart pumps while resting and with different levels of exercise.
* Electrocardiogram (ECG), a test that measures the electrical activity of the heart
* Blood tests

Controls:Blood sample and medical data collected once

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria-Patient

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, any age
* Diagnosed with idiopathic, anorexigen-induced,heritable PAH, PVOD/PCH. Inclusion Criteria-Relative
* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, any age
* Has a family member diagnosed with idiopathic, anorexigen-induced, PVOD/PCH or heritable PAH

Exclusion Criteria-Patient

The participant may not enter the study if ANY of the following apply:

* Patient is unable to give informed consent.
* Not suffering from idiopathic, anorexigen-induced, PVOD/PCH or heritable PAH

Exclusion Criteria-Relative

The participant may not enter the study if ANY of the following apply:

• Patient is unable to give informed consent.

Inclusion criteria-Controls

* Participant is willing and able to give informed consent for participation in the study.
* Self-reported to be healthy
* Age range up to 75 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with idiopathic, anorexigen-induced, heritable PAH or PVOD. Relative who has a family member diagnosed with idiopathic, anorexigen-induced, heritable PAH or PVOD/PCH
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
To recruit a national cohort (1000 subjects) of heritable, idiopathic PAH and PVOD/PCH cases. | 8 years
  The purpose of this study is to set up a national cohort of heritable, idiopathic PAH cases, PVOD/PCH and their relatives, to study the genetic and environmental contributions to disease. Setting up of this cohort of patients and relatives will provide the best resource for understanding what causes or triggers the disease, how to predict risk of death and response to therapy in individual patients, and to provide new ways of preventing and treating pulmonary arterial hypertension. The study will enable a better understanding for the first time the natural history of PAH, whether inherited or not. National outcomes to be measured will include survival, progression of the disease, changes in 6 minute walk distance, admissions to hospital for PAH and cause of death. Incidence of new cases of PAH will be measured in relatives as well.

SECONDARY OUTCOMES:
To recruit PAH patients (1000) and family members to a Biorepository for serum/plasma and urine to identify biomarkers of disease onset, progression and response to treatment. | 8 years
  To establish a Biorepository for serum/plasma, urine, tissues and cells from heritable pulmonary arterial hypertension (HPAH) patients, PVOD/PCH and their relatives, and patients with idiopathic PAH. This will allow studies to identify novel biomarkers of disease onset, progression and response to individual or combination therapies.

OTHER OUTCOMES:
longitudinal clinical evaluation and sampling of HPAH family members | 8 years
  To characterise the natural history of disease onset and progression in the UK national cohort of PAH patients, coupled with longitudinal clinical evaluation and sampling of heritable pulmonary arterial hypertension family members. Longitudinal clinical data will be collated on subjects including haemodynamic data, clinical and research bloods, echocardiographic data, 6 minute walk distance, cardiopulmonary exercise testing, nt-proBNP and safety data ( admissions to hospital PAH related and cause and date of death) and medications.
Elucidation of the underlying genetic architecture of idiopathic and heritable PAH | 8 years
  1000 subjects will have a one off blood sample taken for next generation genetic sequencing (up to their entire genome). Samples will be sequenced to identify novel genetic mutations associated with PAH. A single blood sample will also be taken for mutation testing for BMPR2 and other genes associated with PAH. Outcomes will include identification of novel mutations in PAH

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Morrell, Principal Investigator — University of Cambridge
Locations (8):
- United Kingdom (8):
  - Royal United Hospitals Bath, Bath
  - Royal Papworth Hospital NHS Trust, Cambridge
  - Golden Jubilee National Hospital, Glasgow
  - Imperial Hospital, London
  - Royal Brompton Hospital, London
  - Royal Free Hospital, London
  - Freeman Hospital, Newcastle
  - Sheffield Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No
Consent for sharing of non identifiable study data for regulatory authorities, third parties including commercial companies outside the UK and NHS trusts where it is relevant to taking part in this research.

REFERENCES:
- See also: Study website — http://www.ipahcohort.com
- See also: Pulmonary Hypertension patient website — https://www.phauk.org/